CLINICAL TRIAL: NCT05907616
Title: Feasibility and Impact of the FOOD4MOMS Produce Prescription Program Among Pregnant Latina Women
Acronym: FOOD4MOMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Wholesome Wave (Other); Hispanic Health Council, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000034840
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Food Selection; Food Preferences; Food Insecurity
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pregnant Latina women (Experimental): Pregnant Latina women in Hartford CT enrolled during the first or second trimester of pregnancy. Participants will be provided with up to three nutrition education sessions and will be sent text message reminders to redeem their incentives every month and to provide them with nutrition tips.
  Interventions: Behavioral: Produce purchase incentive

INTERVENTIONS:
Behavioral: Produce purchase incentive — Participants will be provided with a specific incentive amount per month for 10 months to purchase produce, nutrition education sessions and will be sent text message reminders to redeem their incentives every month and to provide them with nutrition tips.

SUMMARY:
The study will include women enrolled during the second trimester of pregnancy who will be provided with a specific amount per month for 10 months to purchase produce. Women will be provided with up to three nutrition education sessions and will be sent text message reminders to redeem their incentives every month and to provide them with nutrition tips. The study will use a co-design approach to utilize feedback from potential participants as well as participants at multiple time points in the process to improve the intervention and make it more relevant and impactful to our population.

DETAILED DESCRIPTION:
This protocol describes the implementation of an intervention to improve access to fruits and vegetables among pregnant Latina women in Hartford CT in partnership with Wholesome Wave of Bridgeport CT, a national leader in nutrition incentive programming and policy.

The target population are pregnant Latina women living in Hartford CT. Having access to the right foods as well as enough food during pregnancy promotes optimal fetal development. A prescription program that provides increased fruit and vegetable access to low-income pregnant women can help improve the diet of women during pregnancy.

Nutrition education sessions (either virtual or in person) will be attended by all participants with one session required and up to two additional sessions optional.

Fruits and vegetables may be purchased at diverse community locations or online for home delivery.

ELIGIBILITY:
Inclusion Criteria:

* during first or second trimester of pregnancy
* live in the city of Hartford
* low income (participating or enrolled in WIC, SNAP or Medicaid)
* speak English or Spanish.

Exclusion Criteria:

* Any individual not meeting any of this criterion will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in amount of produce purchased or accessed | baseline and month 10
  The amount of produce purchased or accessed will be asses using a self-report survey. An increase in produce purchased or accessed indicates a positive outcome.
Change in Produce Intake | baseline and month 10
  Change in Produce Intake will be assessed using a self-report survey. An increase in produce intake indicates a positive outcome.

SECONDARY OUTCOMES:
Change in household food insecurity | baseline and month 10
  Change in household food insecurity assessed using a self-report survey. Less food insecurity indicates a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Pérez-Escamilla, PhD, Principal Investigator — Yale University
Locations (1):
- Hispanic Health Council, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No